CLINICAL TRIAL: NCT06142084
Title: True Ileal Digestibility of Different Plant-based Proteins in a Human Ileostomy Model
Brief Title: Digestibility of Different Plant-based Proteins in Humans With Ileostomy
Acronym: PAN-Prodig
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Dnr 2023-04189-01
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Ileostomy - Stoma
Keywords: Protein; Plant-based; Digestibility
MeSH Terms: interventions — Pea Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dietary Intervention Sequence 1 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 2 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 3 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 4 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 5 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 6 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 7 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 8 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 9 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 10 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal
- Dietary Intervention Sequence 11 (Meals: Pea protein (2x), Oat protein (2x), Protein-free (1x)) (Experimental): The participant will consume the below mentioned meals in a random order on five different study days (one on each visit):
  * Protein meal: pea protein, low bioavailability
  * Protein meal: pea protein, high bioavailability
  * Protein meal: oat protein, low bioavailability
  * Protein meal: oat protein, high bioavailability
  * Protein-free meal
  Interventions: Dietary Supplement: Oat Protein, low bioavailability; Dietary Supplement: Oat Protein, high bioavailability; Dietary Supplement: Pea Protein, low bioavailability; Dietary Supplement: Pea Protein, high bioavailability; Dietary Supplement: Protein-free meal

INTERVENTIONS:
Dietary Supplement: Oat Protein, low bioavailability — Participants will consume a protein meal consisting of cooked whole oat kernels (amount based on body weight, 0.3g of protein/kg bodyweight).
Dietary Supplement: Oat Protein, high bioavailability — Participants will consume a protein meal consisting of heated oat protein concentrate (amount based on body weight, 0.3g of protein/kg bodyweight).
Dietary Supplement: Pea Protein, low bioavailability — Participants will consume a protein meal consisting of cooked whole yellow peas (amount based on body weight, 0.3g of protein/kg bodyweight).
Dietary Supplement: Pea Protein, high bioavailability — Participants will consume a protein meal consisting of heated pea protein isolate (amount based on body weight, 0.3g of protein/kg bodyweight).
Dietary Supplement: Protein-free meal — Participants will consume a protein-free meal to correct analyses for endogenous protein losses.

SUMMARY:
The goal of this interventional study is to learn about the digestibility of different plant-based proteins in adults (age 18-75) with an ileostomy.

The main questions the study aims to answer are:

1. How does the digestibility of proteins in the small intestine differ between different plant-based proteins?
2. Which proteins and amino acids are not digested or absorbed in the small intestine and are available for further metabolic processes in the large intestine?
3. How do metabolites in the collected content of the ileostomy bag differ after consuming different plant-based proteins?
4. Can the in vivo results be compared to results from existing in vitro models?

Participants will consume five different protein meals (oat protein - high bioavailable, oat protein - low bioavailable, pea protein - high bioavailable, pea protein low bioavailable, protein-free meal) on five different study days in a random order. Five hours after consuming the test meals ileostomy bags will be collected and the content will be analysed to answer the above mentioned research questions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 75 years
* Body mass index: 18.5 - 30 kg/m2
* (double-loop) Ileostomy with an intact small bowel
* Signed informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Ileostomy < 3 months before the study
* Any clinically significant present or past disease/condition other than colon cancer which in the investigator's opinion could interfere with the results of the trial
* Any clinically significant present or past medication which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
True ileal digestibility of different plant-based proteins | 0-5 hours after consumption of test meal (on all 5 study days)
  The primary outcome is defined as the differences in the true ileal digestibility, determined by measuring the amount of nitrogen in the meal and the amount of unabsorbed nitrogen in the ileal fluid after consuming four different plant-based protein meals

SECONDARY OUTCOMES:
Protein and metabolite profiles in ileostomy digesta | 0-5 hours after consumption of test meal (on all 5 study days)
  The secondary outcomes are defined as changes in protein and metabolite profiles in the digesta, determined by proteomics and metabolomic analyses.
Differences between in vivo and in vitro data | In vivo data: 0-5 hours after consumption of test meal (on all 5 study days)
  Results from the human ileostomy model will be compared with results from in vitro digestion according to the Infogest 2.0 protocol for each of the tested plant-based proteins

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided